CLINICAL TRIAL: NCT04561063
Title: A Multi-center, Randomised, Open Label Study of Nitazoxanide (NTZ), or Sofosbuvir and Daclatasvir (SOF/DCV), Compared to no Pharmacological Intervention for the Prevention of COVID-19 Disease in Healthcare Workers and Inner City Inhabitants at High Risk of Exposure to SARS-CoV-2
Brief Title: COVID-19 Prophylaxis South Africa (COVER HCW)
Acronym: COVER
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: University of Witwatersrand, South Africa (Other)
Responsible Party: Principal Investigator, Professor Francois Venter, Divisional Director: Ezintsha, University of Witwatersrand, South Africa
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Prevention
Other Study IDs: EZ-SS-025
Record Dates: First submitted 2020-09-21; First posted 2020-09-23 (Actual); Last update posted 2022-06-07 (Actual); Status verified 2022-06

CONDITIONS: Covid19; SARS-CoV Infection
Keywords: Nitazoxanide; Sofosbuvir/Daclatasvir; COVID-19; SARS-CoV-2
MeSH Terms: conditions — COVID-19; Severe Acute Respiratory Syndrome | interventions — nitazoxanide; Sofosbuvir; daclatasvir

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (3):
- Arm A: No pharmacological intervention (PPE only) (No Intervention): No intervention
- Arm B: Nitazoxanide (NTZ) (Active Comparator): Nitozoxanide administered
  Interventions: Drug: Nitazoxanide
- Arm C: Sofosbuvir/daclatasvir (SOF/DCV). (Active Comparator): Sofosbuvir/daclatasvir administered
  Interventions: Drug: Sofosbuvir/Daclatasvir

INTERVENTIONS:
Drug: Nitazoxanide — Nitozoxanide 1 tablet (500 mg) taken 12-hourly with food for the first week, followed by 2 tablets (1000 mg) taken 12-hourly with food thereafter. (Participants that fail to tolerated the 1000 mg 12-hourly dose may revert back to the lower dose.)
  Arms: Arm B: Nitazoxanide (NTZ)
Drug: Sofosbuvir/Daclatasvir — Sofosbuvir/daclatasvir 400mg/60 mg sofosbuvir/daclatasvir fixed dose combination 1 tablet daily
  Arms: Arm C: Sofosbuvir/daclatasvir (SOF/DCV).

SUMMARY:
This is a randomised, multi-center, open label, adaptive, exploratory trial to assess the efficacy of two different drug regimens in terms of preventing symptomatic COVID-19 disease in healthcare workers at high risk of exposure to SARS-CoV-2. The trial will compare two different experimental medication arms to the control arm comprising the use of standard personal protective equipment (PPE) with no additional pharmacological intervention.

DETAILED DESCRIPTION:
This is a randomised, multi-center, open label, adaptive, exploratory trial to assess the efficacy of two different drug regimens in terms of preventing symptomatic COVID-19 disease in healthcare workers at high risk of exposure to SARS-CoV-2. The trial will compare two different experimental medication arms to the control arm comprising the use of standard personal protective equipment (PPE) with no additional pharmacological intervention.

Volunteers will be recruited from participating institutions and community healthcare workers (CHWs) that are responsible for collecting swabs for PCR detection of SARS-CoV-2. Up to 1950 (or 2130 pending funding) eligible participants will be randomised in a 1:1:1 ratio to one of the investigational arms.

Participants will be followed until 65 PCR and serology-confirmed, SARS-CoV-2 infections are identified in the control arm (or 165 in the entire study cohort). For each episode of PCR-confirmed COVID-19 disease, data on self-reported symptoms (modified Flu-PRO) and their duration, and an investigator-assessed severity score (WHO Ordinal Scale for Clinical Improvement) will be recorded. Data on self-reported symptoms and duration will also be collected for other all-cause acute respiratory illnesses. Safety and tolerability of each arm will be assessed through adverse event reporting. Participants who develop COVID-19 disease will have their IMP discontinued but will be followed up in the study until the completion of the trial, where possible. Multiple, discrete occurrences of COVID-19 disease could therefore be identified in a single participant.

Additional arms may be added, or existing ones substituted, should new potential agents be identified or other combinations for prophylaxis be proposed. A formal amendment will be documented should this be considered.

ELIGIBILITY:
Inclusion Criteria:

1. Age ≥18 years of age, inclusive, at the time of signing the informed consent.
2. Willing and able to provide informed consent via an electronic process.
3. Healthcare worker employed at a participating institution that has been identified as high-risk for SARS-CoV-2 exposure (may include doctors, nurses, nurse aids, radiographers, physiotherapists, phlebotomists, technicians, porters, cleaners, laboratory or other personnel identified as being at high risk of exposure), CHW involved in the collection of samples for the identification of SARS-CoV-2 through PCR, and inner city inhabitants at high risk for SARS-CoV-2 exposure due to the nature of their work and frequent use of public transport (may include essential services employees such as fire fighters, law enforcement officers, grocery store employees; and non healthcare workers using public transport at least three times a week).
4. Women of reproductive potential must be using a highly effective method of contraception prior to enrolment or must be willing to start a method at enrolment and continue its use throughout the duration of the study.
5. Body weight ≥45 kg.
6. Access to reliable video conference, telephone, direct/text messaging, or other device permitting real-time, reliable information transfer.

Exclusion Criteria:

1. Pregnant or lactating women.
2. PCR and/or serology confirmed SARS-Cov-2 infection at screening.
3. Current symptoms of COVID-19 disease (including, but not limited to, fever or chills, cough, myalgia, sore throat, shortness of breath, or new onset of anosmia or ageusia, or diarrhea).
4. Self-reported presence or history of any of the following conditions:

   * Chronic kidney disease (Stage IV or receiving dialysis)
   * Cirrhosis (Child-Pugh Class B or greater)
   * Porphyria cutanea tarda.
5. Currently on treatment for epilepsy or other seizure disorder.
6. Currently on treatment with a protease inhibitor-based antiretroviral regimen, or efavirenz, or on treatment with amiodarone, carbamazepine, phenobarbitone, phenytoin, primidone, rifampicin,St. John's wort or any herbal products which may potentially decrease the concentration of the IMP.
7. Known hypersensitivity or specific contraindications to the use of any of the active drugs in the treatment arms or similar compounds.
8. Current enrolment in another COVID-19 prevention trial.
9. History of alcohol abuse within the last 6 months.
10. Having history or have risk factors for brady-arrhythmias (those with undiagnosed cardiac conditions).
11. History of malignancies in the last 5 years, excluding in-situ or non-invasive malignancies.
12. Concurrent or recent (within 3 months) participation in other research with a compound likely to interfere with any of the investigational products.
13. Any surgical or medical condition which might significantly alter the absorption, distribution, metabolism, or excretion of drugs, or which may jeopardize the safety of the volunteer or the objectives of the study. The Investigator should make this determination in consideration of the volunteer's medical history.
14. Inability or unwillingness to be followed up for the study period.
15. Personnel (e.g. investigator, sub-investigator, research assistant, pharmacist, study coordinator or anyone mentioned in the delegation log) directly involved in the conduct of the study. (Personnel employed at a study site, but not directly involved in the conduct of the study, who would like to participate in the study, may only do so if they are enrolled in the study through a different site at which they are not employed.)
16. Participant is judged by the Investigator to be at significant risk of failing to comply with the provisions of the protocol as to cause harm to self or seriously interfere with the validity of the study results.
17. Confirmed vaccination against SARS-Cov-2.

Ages: 18 Years to 99 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 1950 (Actual)
Dates: Start 2020-12-08 (Actual); Primary Completion 2022-02-28 (Actual); Study Completion 2022-02-28 (Actual)

PRIMARY OUTCOMES:
Number of SARS-CoV-2 infections | 6 months
  Number of SARS-CoV-2 infection (COVID-19) confirmed by PCR and/or serology.

SECONDARY OUTCOMES:
Duration of symptoms | 6 months
  Duration of symptoms for each symptomatic infection
Maximum score on WHO Ordinal Scale | 6 months
  Maximum score on WHO Ordinal Scale for Clinical Improvement for each symptomatic infection. Score of 0 being uninfected and a score of 8 being dead.
Time to onset of SARS-CoV-2 infection | 6 months
  Time to onset of SARS-CoV-2 infection (COVID-19) confirmed by PCR and/or serology
Number of symptomatic SARS-CoV-2 infections | 6 months
  Number of symptomatic SARS-CoV-2 infection (COVID-19) confirmed by PCR and/or serology
Number of asymptomatic SARS-CoV-2 infections | 6 months
  Number of asymptomatic • Asymptomatic SARS-CoV-2 infection suggested by serological outcome
Peak score on modified Flu PRO | 6 months
  Peak score on modified Flu-PRO during each symptomatic infection. 37-item questionairre assessing the severity of flu like symptoms one a scale of 0 - not at all to 5 - very much.

CONTACTS AND LOCATIONS:
Overall Officials: Simiso Sokhela, Principal Investigator — Ezintsha
Locations (2):
- South Africa (2):
  - Charlotte Maxeke Johannesburg Academic Hospital, Johannesburg, Gauteng
  - Sunnyside Office Park, Johannesburg, Gauteng

REFERENCES:
- [Derived] Kreuzberger N, Hirsch C, Chai KL, Tomlinson E, Khosravi Z, Popp M, Neidhardt M, Piechotta V, Salomon S, Valk SJ, Monsef I, Schmaderer C, Wood EM, So-Osman C, Roberts DJ, McQuilten Z, Estcourt LJ, Skoetz N. SARS-CoV-2-neutralising monoclonal antibodies for treatment of COVID-19. Cochrane Database Syst Rev. 2021 Sep 2;9(9):CD013825. doi: 10.1002/14651858.CD013825.pub2. PMID 34473343